CLINICAL TRIAL: NCT01462747
Title: An Open Prospective Study Evaluating the Efficacy and Safety of a Medical Device,KULIST, for the Treatment of Chronic, Non-complicated Perianal Fistulas
Brief Title: Efficacy and Safety Study of a Medical Device (KULIST)to Treat Perianal Fistulas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nordic Drugs AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KULIST-001
Record Dates: First submitted 2011-10-21; First posted 2011-10-31 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Perianal Fistulas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KULIST (Experimental): Medical Device, Activated carbon
  Interventions: Device: KULIST

INTERVENTIONS:
Device: KULIST — Twice daily dosing for 8 weeks

SUMMARY:
The aim of this study is to evaluate the effects of rectally administered activated carbon (medical device KULIST) in chronic, uncomplicated, perianal fistulas.

DETAILED DESCRIPTION:
Patients with chronic uncomplicated perianal fistulas located below levator ani will be treated twice daily with KULIST for 8 weeks. The efficacy will be evaluated by means of an overall clinical evaluation of fistula closure, as well as by anal ultrasonography.

Also changes in Patient Assessment of Symptoms and Impact on Daily Function will be evaluated. Safety will be evaluated by standard adverse event /adverse device effects reporting.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with perianal fistulas diagnosed by clinical examination and evaluated as "not healed/open"
2. Fistula classified as intersphincteric and transsphincteric according to Parks´classification (Parks 1976)
3. Superficial fistula involving a part of the external sphincter muscle
4. Age: ≥18 years and ≤ 75 years
5. Informed consent and/or Letter of Authority (as applicable) obtained

   Exclusion Criteria
6. Inflammatory Bowel Disease (IBD)
7. Rectovaginal fistulas
8. Rectourethral fistulas
9. Rectovesical fistulas
10. Extra-sphincteric and supra-sphincteric fistula according to Parks´classification
11. Complicated fistulas (eg. horse shoe fistulas) as evaluated by the investigator.
12. Any surgical treatment for perianal fistulas
13. Colorectal and/or anal malignancy
14. Other malignancy requiring active treatment
15. Subcutaneous fistulas not involving any part of the external sphincter
16. Other diseases which as per the investigator's opinion should be contraindicated
17. Subjects who are not able to complete study procedures as per the investigator's opinion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of fistula healing, change from baseline | week 8 and 24
  Fistula assessed as healed/not healed

SECONDARY OUTCOMES:
Anal ultrasonography, change from baseline | week 8 and 24
  Healed/not healed
Patient assessment of Symptoms and Impact on Daily Function, change from baseline | week 8 and 24
  By the use of VAS scales and questionnaires the patients subjective evaluations of symptoms and impact on daily living will be assessed
Safety, change from baseline | week 2, 8, 24
  Standard collection of adverse events and adverse device effects.

CONTACTS AND LOCATIONS:
Overall Officials: Måns Bohe, MD, PhD, Principal Investigator — Skane University Hospital
Locations (2):
- Sweden (2):
  - Malmö University Hospital Dept of Surgery, Malmo, Malmö
  - Kolorektalsektionen Kirurg -och urologkliniken Danderyds Sjukhus AB, Stockholm, Stockholm County